CLINICAL TRIAL: NCT06773104
Title: Autogenous Tooth Bone Graft Versus Allogeneic Bone Graft Around Dental Implant in Aesthetic Zone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Diab Abdel Gaied Diab Ghanem Mohammed, principal investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: diab123
Record Dates: First submitted 2024-12-30; First posted 2025-01-14 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Immediate Dental Implants; Thin Labial Plate of Bone Pre-extraction; Hopeless Tooth in Esthetic Zone
Keywords: autogenous tooth bone graft; allogenic bone graft; grafting the jumbing gap; immediate dental implant

STUDY DESIGN:
Intervention Model Description: non restorable anterior teeth with thin labial plate of bone
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autogenous tooth bone graft group (Experimental): Twelve patients receiving immediate implant placement with autogenous fresh partially demineralized dentin graft.
  Interventions: Procedure: Allogeneic bone graft with immediate implant placement
- Allogeneic bone graft group (control group) (Active Comparator): Patients receiving immediate dental implant placement with allogeneic bone graft (DFDBA) for grafting of the jumping gap.
  Interventions: Procedure: immediate implant with allogenic bone graft

INTERVENTIONS:
Procedure: immediate implant with allogenic bone graft — after atraumatic extraction immediate implant will be inserted with allogenic bone graft
  Arms: Allogeneic bone graft group (control group)
Procedure: Allogeneic bone graft with immediate implant placement — Immediate dental implant placement with grafting of the jumping gap using allogeneic bone graft (DFDBA).
  Arms: Autogenous tooth bone graft group

SUMMARY:
24 patienta with non restorable anterior teeth underwent extraction with immediate implant installation using bone grafts either autogenous tooth bone graft or allogenic bone graft Autogenous tooth bone graft group (study group): 12 patients will have immediate implant placement with autogenous tooth bone graft.

• Allogeneic bone graft group (control group): 12 patients will have immediate implant placement with allogeneic bone graft (demineralized freeze dried bone allograft - cortico cancellous).

DETAILED DESCRIPTION:
24 patienta with non restorable anterior teeth underwent extraction with immediate implant installation randomized to two groups Autogenous tooth bone graft group (study group): 12 patients will have immediate implant placement with autogenous tooth bone graft.

• Allogeneic bone graft group (control group): 12 patients will have immediate implant placement with allogeneic bone graft (demineralized freeze dried bone allograft - cortico cancellous).

preparation of autogenous tooth bone graft Any restorations, caries, cementum, periodontal ligament and pulp tissue will be removed .The tooth will be grinded using dental bone mill and bone crusher Tooth particles will be sieved to particles size 300 to 1200 microns. The sorted particles will be immersed in 70 % ethanol and 5% Peracetic acid* in a sterile container for 10 minutes to remove any soft tissue remnants, bacteria and smear layer (defatting and sterilization).

Tooth particles will be demineralized using 2% HNO3for 20 minutes to expose the dentine organic matrix.

The bacteria-free particulate dentin will be washed with phosphate buffered saline‡ twice for 5 minutes to restore the PH balance to 7.4. In the same setting, surgical procedure after atraumatic extraction immediate implant willbe inserted according to dimensions taken from CBCT and jumbing gap will be filled with bone graft according to randomization

ELIGIBILITY:
Inclusion Criteria:

Patients with non restorable maxillary anterior teeth need to be extracted.

* Thin labial plate of bone of the tooth to be extracted.
* Patients age above 20years old.
* Good oral hygiene.
* No signs of acute infection or inflammation

Exclusion Criteria:

* Prior radiation therapy.
* Soft and hard tissue pathology at the operation site.
* Any relevant systemic disease or medication that might compromise bone healing.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-03-25 (Actual); Primary Completion 2025-10-16 (Actual); Study Completion 2025-10-16 (Actual)

PRIMARY OUTCOMES:
labial bone thickness | 6 months
  measuring thickness of labial bone labial to the implant
marginal bone loss | 6 months

SECONDARY OUTCOMES:
bone density around dental implant | 6 months
  bone density will be assessed using CBCT buccal to the implant fixtures 6 months after implant installation
implant secondary stability | 6 months
  Implant stability will be assessed at the time of implant insertion and 6 months after the operation. Resonance frequency analysis (RFA) values expressed as implant stability quotient (ISQ) will be recorded by a transducer attached to the implant by a screw and a frequencyresponse analyzer (Osstell Mentor Device) with the average of 2measurements performed with the probe in 2 perpendiculardirections
implant success | 6 months
  when the following clinical features arise: emerging of the fistula, the particle of the bone graft material flow out from the fistula or mucosal dehiscence, and the chronic inflammation ragarded as failure

CONTACTS AND LOCATIONS:
Overall Officials: diab abdelgaied diab, master, Principal Investigator — faculty of dentistry tanta university; Rafic ramadan bedir, professor, Principal Investigator — faculty of dentistry tanta university; Ibrahim mohammed nowair, professor, Principal Investigator — faculty of dentistry tanta university; Mona samy sheta, lecturer, Principal Investigator — faculty of dentistry tanta university
Locations (1):
- Faculty of Dentistry, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No